CLINICAL TRIAL: NCT06643559
Title: Investigating The Effect Of Cognitive Rehabilitation On Cognitive Impairment Associated With Antiseizure Medications In Patients With Epilepsy
Brief Title: The Effect of Cognitive Rehabilitation on Epileptic Pateints Under Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Omer Karadas, Prof.Dr.Omer Karadas, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR ethics commitee 2022/84
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Dysfunction; Epilepsy
Keywords: cognitive rehabillitation; antiseizure medication; MoCA; P300, N200
MeSH Terms: conditions — Cognitive Dysfunction; Epilepsy | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Before monotherapy, newly diagnosed epileptic patients evaluted by MoCA and P300. The patients began their treatments, and from the next day, computer-based cognitive rehabilitation was randomly assigned to some patients in each drug group, four times a week. For each drug, patients were randomly divided into those who did not receive (A) and those who received (B) cognitive rehabilitation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with cognitive rehabilitation (Active Comparator): Patient which have started antiseizure monotherapy plus have been included cognitive rehabilitation programme.
  Interventions: Other: cognitive rehabilitation
- Patients Without Cognıtıve Rehabilitation (No Intervention)

INTERVENTIONS:
Other: cognitive rehabilitation — Cognitive rehabilitation started to one group at the beginning of the antiseizure medicine. Participants underwent computer-based cognitive rehabilitation for 3 sessions per week, with each session lasting an average of 60 minutes. Before the sessions, all participants were given detailed information about the programme and its use. The rehabilitation process was carried out in three areas of cognitive functions: memory, executive functions, and language skills.
  Arms: patients with cognitive rehabilitation

SUMMARY:
It is clear that studies on cognitive rehabilitation in epilepsy patients mostly focus on patients undergoing epilepsy surgery and are largely classified according to the type of epilepsy. The main purpose of this study is to determine whether cognitive impairments associated with antiepileptic drugs develop in epilepsy patients using neuropsychological tests and event-related potentials, and if such an impairment is present, to investigate whether cognitive rehabilitation is beneficial.

DETAILED DESCRIPTION:
Patients who were planned to start monotherapy were first included in the study by performing a face-to-face MoCA test. After the MoCA test, experienced neurologists measured event-related potentials, including P300 and N200 potentials and N2P3 amplitudes, in the electrophysiology laboratory. Patients for each drug were randomly assigned to the no cognitive rehabilitation group (A) or the cognitive rehabilitation group (B). At the end of the second month, MoCA test and event-related potential measurements were performed again in both groups, and the results were analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of epilepsy, -
* Before monotherapy had started

Exclusion Criteria:

* diagnosis of psychogenic non-epileptic seizures,
* epileptic patients currently receiving antiepileptic drugs,
* epileptic patients exhibiting cognitive dysfunction
* epileptic patientswith dementia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 368 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
MoCA | 2 months
  The Montreal Cognitive Assessment (MoCA) is a 30-point screening test that takes approximately 10 minutes to administer. It assesses executive functioning, visuospatial abilities, memory, attention, working memory, language, and orientation. It has high sensitivity and specificity. the maximum score is 30. Higher scores mean a better outcome.
Cognitive Event Related Potentials | 2 months
  The standardized recording protocol was utilized to acquire reliable and consistent Event-Related Potentials (ERP) data for a comprehensive evaluation of the brain's response to auditory stimuli. In the analysis of potentials, the amplitude between the N200 and P300 was measured from the N200 peak to the P300 peak. The latencies of the N200 and P300 potentials were also determined by identifying the midpoint of each potential (latencies in miliseconds (ms) and amplitudes in microvolt (uV))

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Reseach Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Baxendale S. Cognitive rehabilitation and prehabilitation in people with epilepsy. Epilepsy Behav. 2020 May;106:107027. doi: 10.1016/j.yebeh.2020.107027. Epub 2020 Mar 21. PMID 32208338
- [Result] Choi J, Twamley EW. Cognitive rehabilitation therapies for Alzheimer's disease: a review of methods to improve treatment engagement and self-efficacy. Neuropsychol Rev. 2013 Mar;23(1):48-62. doi: 10.1007/s11065-013-9227-4. Epub 2013 Feb 12. PMID 23400790
- [Result] Duncan CC, Barry RJ, Connolly JF, Fischer C, Michie PT, Naatanen R, Polich J, Reinvang I, Van Petten C. Event-related potentials in clinical research: guidelines for eliciting, recording, and quantifying mismatch negativity, P300, and N400. Clin Neurophysiol. 2009 Nov;120(11):1883-1908. doi: 10.1016/j.clinph.2009.07.045. Epub 2009 Sep 30. PMID 19796989
- [Result] Farina E, Raglio A, Giovagnoli AR. Cognitive rehabilitation in epilepsy: An evidence-based review. Epilepsy Res. 2015 Jan;109:210-8. doi: 10.1016/j.eplepsyres.2014.10.017. Epub 2014 Nov 6. PMID 25524861
- [Result] Ismail Z, Aguera-Ortiz L, Brodaty H, Cieslak A, Cummings J, Fischer CE, Gauthier S, Geda YE, Herrmann N, Kanji J, Lanctot KL, Miller DS, Mortby ME, Onyike CU, Rosenberg PB, Smith EE, Smith GS, Sultzer DL, Lyketsos C; NPS Professional Interest Area of the International Society of to Advance Alzheimer's Research and Treatment (NPS-PIA of ISTAART). The Mild Behavioral Impairment Checklist (MBI-C): A Rating Scale for Neuropsychiatric Symptoms in Pre-Dementia Populations. J Alzheimers Dis. 2017;56(3):929-938. doi: 10.3233/JAD-160979. PMID 28059789
- [Result] Ismail Z, Rajji TK, Shulman KI. Brief cognitive screening instruments: an update. Int J Geriatr Psychiatry. 2010 Feb;25(2):111-20. doi: 10.1002/gps.2306. PMID 19582756
- [Result] Engelberts NH, Klein M, Ader HJ, Heimans JJ, Trenite DG, van der Ploeg HM. The effectiveness of cognitive rehabilitation for attention deficits in focal seizures: a randomized controlled study. Epilepsia. 2002 Jun;43(6):587-95. doi: 10.1046/j.1528-1157.2002.29401.x. PMID 12060017
- [Result] Jones MK. Imagery as a mnemonic aid after left temporal lobectomy: contrast between material-specific and generalized memory disorders. Neuropsychologia. 1974 Jan;12(1):21-30. doi: 10.1016/0028-3932(74)90023-2. No abstract available. PMID 4821186
- [Result] Koorenhof L, Baxendale S, Smith N, Thompson P. Memory rehabilitation and brain training for surgical temporal lobe epilepsy patients: a preliminary report. Seizure. 2012 Apr;21(3):178-82. doi: 10.1016/j.seizure.2011.12.001. Epub 2011 Dec 23. PMID 22197200
- [Result] Loring DW, Meador KJ. Epilepsy: maximizing cognitive outcomes in epilepsy. Nat Rev Neurol. 2012 Aug;8(8):416-7. doi: 10.1038/nrneurol.2012.143. Epub 2012 Jul 10. No abstract available. PMID 22777245
- [Result] Ortinski P, Meador KJ. Cognitive side effects of antiepileptic drugs. Epilepsy Behav. 2004 Feb;5 Suppl 1:S60-5. doi: 10.1016/j.yebeh.2003.11.008. PMID 14725848
- [Result] Ponds RW, Hendriks M. Cognitive rehabilitation of memory problems in patients with epilepsy. Seizure. 2006 Jun;15(4):267-73. doi: 10.1016/j.seizure.2006.02.011. Epub 2006 Mar 23. PMID 16563809
- [Result] Quon RJ, Mazanec MT, Schmidt SS, Andrew AS, Roth RM, MacKenzie TA, Sajatovic M, Spruill T, Jobst BC. Antiepileptic drug effects on subjective and objective cognition. Epilepsy Behav. 2020 Mar;104(Pt A):106906. doi: 10.1016/j.yebeh.2020.106906. Epub 2020 Jan 29. PMID 32006792
- [Result] Rosca EC, Simu M. Montreal cognitive assessment for evaluating cognitive impairment in multiple sclerosis: a systematic review. Acta Neurol Belg. 2020 Dec;120(6):1307-1321. doi: 10.1007/s13760-020-01509-w. Epub 2020 Sep 29. PMID 32996098
- [Result] Shafiyev J, Karadas O. The assessment of the impact of antiepileptic drugs on cognitive functions via N-200/P-300 potentials and neuropsychological measures. Neurol Sci. 2024 Oct;45(10):5011-5021. doi: 10.1007/s10072-024-07606-5. Epub 2024 May 25. PMID 38795272
- [Result] Witt JA, Elger CE, Helmstaedter C. Adverse cognitive effects of antiepileptic pharmacotherapy: Each additional drug matters. Eur Neuropsychopharmacol. 2015 Nov;25(11):1954-9. doi: 10.1016/j.euroneuro.2015.07.027. Epub 2015 Aug 6. PMID 26296280
- [Result] Witt JA, Helmstaedter C. Cognition in the early stages of adult epilepsy. Seizure. 2015 Mar;26:65-8. doi: 10.1016/j.seizure.2015.01.018. Epub 2015 Feb 7. PMID 25799904